CLINICAL TRIAL: NCT01117051
Title: A 12-week, Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Prucalopride in Subjects With Chronic Non-cancer Pain Suffering From Opioid Induced Constipation
Brief Title: Prucalopride Effects on Subjects With Chronic Non-cancer Pain Suffering From Opioid Induced Constipation
Acronym: OIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped by the sponsor based on a non-safety related business priority decision
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M0001-C301; SPD555-301 (Other: Shire Development LLC); 2009-015652-20 (EudraCT Number)
Record Dates: First submitted 2010-04-29; First posted 2010-05-05 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Non-cancer Pain; Opioid Induced Constipation
Keywords: Opioid induced constipation/prucalopride chronic non-cancer pain; Subjects with chronic non-cancer pain suffering from OIC
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- Resolor (Active Comparator): prucalopride
  Interventions: Drug: prucalopride

INTERVENTIONS:
Drug: placebo — placebo
  Arms: placebo
Drug: prucalopride — 1 or 2 mg prucalopride once daily before breakfast
  Arms: Resolor

SUMMARY:
The study will evaluate the efficacy, safety and tolerability of prucalopride over 12 weeks of treatment in subjects aged 18 years and older with chronic non-cancer pain, suffering from opioid induced constipation.

ELIGIBILITY:
Inclusion criteria to be assessed at screening:

1. Male or non-pregnant, non-breast-feeding female outpatient ≥18 years.
2. Has chronic pain of any aetiology (except cancer pain) requiring daily maintenance treatment with opioids;has been on stable daily opioid dose during at least the previous 2 weeks; and is expected to remain on stable daily dose of opioids for at least 15 weeks after Visit 1.
3. Subject is suffering from OIC (i.e. secondary to chronic opioid use).
4. Subject agrees to stop his/her laxative treatment and is willing to use rescue medication.

Main exclusion criteria to be assessed at screening:

1. Constipation is thought to be drug-induced (except for opioids)
2. Disallowed medication is being used
3. Subject was on chronic therapy for chronic constipation prior to start of opioid therapy
4. Subject is suffering from secondary causes of chronic constipation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2012-08-13 (Actual); Study Completion 2012-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Leuven, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo once daily before breakfast for up to 12 weeks
- Prucalopride: 1 or 2 mg prucalopride once daily before breakfast for up to 12 weeks
Period: Overall Study
Arm/Group | Placebo | Prucalopride
Started | 86 | 88
Completed | 73 | 77
Not Completed | 13 | 11
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Adverse Event | 4 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not meet in-/exclusion criteria | 0 | 1
Not completed — Sponsor's decision | 3 | 1
Not completed — Surgical procedure | 0 | 1
Not completed — Randomized by mistake | 0 | 1
Not completed — Convenience issue | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population was used which includes all subjects who were randomized into the study and who had received at least 1 dose of investigational product. 174 subjects were randomized but 5 were not treated (n = 169).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Prucalopride | Total
Number analyzed (Participants) | 83 | 86 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (11.67) | 55.7 (12.15) | 56.7 (11.92)
Age, Customized [Count of Participants; unit: Participants]
  Between >=18 and <65 years | 62 | 66 | 128
  Between >=65 and <75 years | 11 | 11 | 22
  >=75 years | 10 | 9 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 62 | 123
  Male | 22 | 24 | 46
Region of Enrollment [Count of Participants; unit: Participants] — All randomized subjects (n = 174)
  Participants
    Belgium | 8 | 9 | 17
    Bulgaria | 4 | 5 | 9
    Czech Republic | 40 | 38 | 78
    Germany | 6 | 7 | 13
    France | 2 | 2 | 4
    United Kingdom | 13 | 14 | 27
    Hungary | 2 | 1 | 3
    Netherlands | 0 | 1 | 1
    Poland | 6 | 5 | 11
    Romania | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With an Average Frequency of >=3 Spontaneous Bowel Movements Per Week
Description: A bowel movement (BM) was defined as spontaneous if no laxatives were taken in the 24 hours preceding that BM.
Time Frame: 12 weeks
Population: Intent-to-Treat (ITT) population includes all subjects who were randomized into the study and who had received at least 1 dose of investigational medication.
Measure: Number; unit: percentage of subjects
Groups:
- Placebo: once daily before breakfast for up to 12 weeks
Arm/Group | Placebo | Prucalopride
Number analyzed (Participants) | 83 | 86
percentage of subjects | 39.8 | 48.8
Statistical Analysis 1: Comparison: Placebo vs Prucalopride; Test type: Superiority or Other; p = 0.305, Cochran-Mantel-Haenszel

2. Secondary Outcome: Plasma Concentration of Prucalopride at Week 2
Time Frame: Week 2
Population: ITT (subjects in the ITT whose post-dose samples were collected outside the 5-hour sampling window were not used in the plasma concentration calculation)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Prucalopride
Number analyzed (Participants) | 62
ng/ml
  pre-dose | 2.827 (1.5989)
  5 hours post-dose | 6.107 (2.8839)

3. Secondary Outcome: Plasma Concentration of Prucalopride at Week 8
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Prucalopride
Number analyzed (Participants) | 53
ng/ml
  pre-dose | 3.179 (1.9066)
  5 hours post-dose | 6.615 (2.5758)

ADVERSE EVENTS:
Arm/Group | Placebo | Prucalopride
Serious Adverse Events (participants affected / at risk) | 2/83 | 2/86
Other Adverse Events (participants affected / at risk) | 30/83 | 30/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | Prucalopride (N=86)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=83) | Prucalopride (N=86)
Nausea (Gastrointestinal disorders) | 5 | 9
Flatulence (Gastrointestinal disorders) | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Influenza (Infections and infestations) | 1 | 2
Headache (Nervous system disorders) | 2 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.